CLINICAL TRIAL: NCT01903954
Title: A Phase 2, Randomized, Double-Blind, Placebo-Controlled Trial of the Safety and Efficacy of ANA598 Administered With Pegylated Interferon and Ribavirin in Genotype 1 Patients With Chronic Hepatitis C Infection
Brief Title: A Study of Setrobuvir in Combination With Pegasys (Peginterferon Alfa-2a) and Copegus (Ribavirin) in Patients With Genotype 1 Chronic Hepatitis C
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NP28302; NCT01281423 (obsolete NCT alias)
Record Dates: First submitted 2013-07-17; First posted 2013-07-19 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Hepatitis C, Chronic
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — peginterferon alfa-2a; Ribavirin; setrobuvir

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Active Comparator (Active Comparator): Pplacebo in combination with standard of care Pegasys (peginterferon alfa-2a) and Copegus (ribavirin)
  Interventions: Drug: peginterferon alfa-2a [Pegasys]; Drug: placebo; Drug: ribavirin [Copegus]
- Setrobuvir (Experimental): Setrobuvir (800 mg orally b.i.d loading dose followed by 200 mg orally .b.i.d.) in combination with standard of care Pegasys (peginterferon alfa-2a) and Copegus (ribavirin)
  Interventions: Drug: peginterferon alfa-2a [Pegasys]; Drug: ribavirin [Copegus]; Drug: setrobuvir

INTERVENTIONS:
Drug: peginterferon alfa-2a [Pegasys] — 180 mcg sc weekly
Drug: placebo — Orally b.i.d.
  Arms: Active Comparator
Drug: ribavirin [Copegus] — 1000 mg or 1200 mg orally daily
Drug: setrobuvir — Loading dose of 800 mg orally b.i.d on Day 1, followed by 200 mg orally b.i.d., 28 or 48 weeks
  Other Names: ANA598
  Arms: Setrobuvir

SUMMARY:
This randomized, double-blind, placebo-controlled study will evaluate the efficacy and safety of setrobuvir in patients with genotype 1 chronic hepatitis C. Treatment-naïve patients will be randomized to receive either setrobuvir (800 mg orally b.i.d loading dose followed by 200 mg orally .b.i.d.) or placebo in combination with standard of care Pegasys (peginterferon alfa-2a) and Copegus (ribavirin). Treatment duration will be 28 weeks or 48 weeks depending on response. Treatment-experienced patients categorized as relapsers, partial responders and viral breakthrough patients to previous pegylated interferon and ribavirin therapy will be randomized to receive either setrobuvir or placebo in combination with Pegasys and Copegus for 48 weeks. Treatment-experienced patients categorized as null-responders to previous pegylated interferon and ribavirin therapy will be assigned to treatment with setrobuvir plus Pegasys and Copegus for 48 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, 18 to 65 years of age inclusive
* Documented chronic hepatitis C
* Treatment-naïve (no prior exposure to Pegasys, Copegus, or experimental HCV therapy) or treatment-experienced with current standard of care (Pegasys and Copegus) but categorized as null-responder or patients with partial response, relapse or viral breakthrough during or following prior treatment
* Serum HCV RNA >/= 50,000 IU/mL at screening
* HCV antibody positive at screening
* HCV genotype 1
* Body mass index (BMI) 18-38 kg/m2
* In good health other than chronic HCV infection in the judgment of the principal investigators
* Negative for hepatitis B and HIV infection

Exclusion Criteria:

* Pregnant or breastfeeding women
* For treatment-naïve patients: any previous treatment for HCV infection
* For treatment-experienced patients: previous treatment with an experimental therapy for HCV infection
* Co-infection with HIV or hepatitis C virus (HBV)
* History or evidence of decompensated liver disease
* History or evidence of hepatocellular carcinoma
* History of alcohol abuse and/or other drug addiction </= 1 year prior to enrollment in the study
* Poorly controlled diabetes mellitus
* One or more additional known primary causes of liver disease other than hepatitis C
* History of acute or chronic pancreatitis
* Participation in an other clinical study of a new chemical entity within 30 days prior to study randomization

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 283 (Actual)
Dates: Start 2011-01; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Proportion of patients achieving sustained virologic response (SVR24), defined as undetectable hepatitis C virus (HCV) RNA at 24 weeks after discontinuation of all study drugs | 24 weeks after discontinuation of all study drugs (treatment duration 28 or 48 weeks)

SECONDARY OUTCOMES:
Proportion of patients achieving undetectable HCV RNA (defined as HCV RNA < 15 IU/mL) at each visit through Week 24 | 24 weeks
Proportion of treatment-naïve patients eligible to stop all treatment at Week 28 | 28 weeks
Safety: Incidence of adverse events | up to approximately 72 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche